CLINICAL TRIAL: NCT06472869
Title: Assessing E-Cigarettes for Tobacco Harm Reduction in the Context of Lung Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024p001502
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Electronic Cigarette Use; Smoking, Cigarette; Nicotine Dependence
Keywords: Tobacco Use Disorder
MeSH Terms: conditions — Vaping; Cigarette Smoking; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Open-label single-arm pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NJOY ACE e-cigarette provision (Experimental): Device: NJOY ACE e-cigarette, 5% nicotine in tobacco flavor
  Patients will be provided with a NJOY ACE electronic cigarette for 4 weeks and asked to use the NJOY ACE as a substitute for smoking combustible cigarettes during the 4 weeks.
  Interventions: Other: NJOY ACE e-cigarette

INTERVENTIONS:
Other: NJOY ACE e-cigarette — Patients will be provided with NJOY ACE electronic cigarettes and 5% nicotine e-liquid cartridges in tobacco flavor for 4 weeks and asked to use the electronic cigarette as a substitute for smoking combustible cigarettes during the 4 weeks

SUMMARY:
This study investigates the feasibility, acceptability, and short-term effects of providing 4 weeks of complimentary electronic cigarettes (ECs) to 30 individuals who did not quit after smoking cessation treatment provided in the context of lung cancer screening and do not plan to quit smoking. This open-label single-arm pilot clinical trial will test the impact of EC provision on: 1) study feasibility, 2) EC acceptability, 3) tobacco use behavior (e.g., cigarettes per day, EC use), and 4) biomarkers (e.g., carbon monoxide, cotinine, and anabasine). Participants will be asked to switch from combustible cigarettes to the NJOY ACE 5% nicotine electronic cigarette (EC) for 4 weeks. They will be followed an additional 4 weeks after EC provision ends (to 8 weeks).

The first study hypothesis is that more than 40% of eligible smokers who are offered participation in the trial will enroll, and that 75% of enrollees will complete the trial. The second study hypothesis is that participants will report fewer cigarettes smoked per day at the end of 4 weeks of EC provision, relative to their baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Participants who completed the Screen Assist study (NCT03611881) and self-reported smoking cigarettes at the end of the study were asked to complete a survey to ascertain their potential interest in participating in a research study to test the effects of switching from combustible cigarettes (CC) to electronic cigarettes (EC). Individuals who expressed interest in switching to EC on that survey were screened for eligibility for this pilot study
* Smoked ≥5 cigarettes/day in past month
* Smoking status at study entry confirmed by breath carbon monoxide (CO) ≥ 6ppm
* Willing to try switching from CC to EC for 4 weeks
* Owns a mobile telephone
* English speaking
* Willing to travel to the Massachusetts General Hospital campus for 3 in-person visits.

Exclusion Criteria:

* Plans to quit smoking and has set a quit date in the next 30 days
* Used smoking cessation treatment in the past 30 days
* Used EC on >2 days in the past 30 days
* Hospitalized for acute coronary syndrome, unstable angina, congestive heart failure, stroke, pneumonia or chronic pulmonary disease/asthma exacerbation in the past 1 month
* Not willing to abstain from smoking marijuana in the 24h before each study visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A. Rigotti, MD, Principal Investigator — Massachusetts General Hospital; Jaqueline C Avila, PhD, Principal Investigator — University of Massachusetts, Boston
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NJOY ACE E-cigarette Provision: Device: NJOY ACE e-cigarette, 5% nicotine in tobacco flavor
  Patients will be provided with a NJOY ACE electronic cigarette for 4 weeks and asked to use the NJOY ACE as a substitute for smoking combustible cigarettes during the 4 weeks.
  NJOY ACE e-cigarette: Patients will be provided with NJOY ACE electronic cigarettes and 5% nicotine e-liquid cartridges in tobacco flavor for 4 weeks and asked to use the electronic cigarette as a substitute for smoking combustible cigarettes during the 4 weeks
Period: Overall Study
Arm/Group | NJOY ACE E-cigarette Provision
Started | 15
Completed (Week 4 Primary Outcome Visit) | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NJOY ACE E-cigarette Provision
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 13
  Non-Hispanic Other | 1
  Hispanic | 1
Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: cigarettes/day] | 16.9 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility
Description: Participant enrollment, measured by the proportion of eligible participants who enroll in the study. Retention is measured by weeks of study participation.
Time Frame: 4 weeks
Population: The number of participants analyzed is different than the sample size as the outcome is participant enrollment among those eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | NJOY ACE E-cigarette Provision
Number analyzed (Participants) | 28
Participants | 15

2. Primary Outcome: Cigarettes Per Day (CPD) Smoked During the Period of E-cigarette Provision
Description: Change in self-reported CPD smoked in the past week assessed using timeline follow-back (TLFB) between baseline and end of e-cigarette provision (Baseline vs.Week 4)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | NJOY ACE E-cigarette Provision
Number analyzed (Participants) | 15
cigarettes/day
  Baseline | 16.9 (7.0)
  Week 4 | 10.2 (7.0)

3. Secondary Outcome: Carbon Monoxide (CO) Concentration in Expired Air
Description: Change in participant's expired air carbon monoxide (CO) concentration assessed via Smokerlyzer during the period of e-cigarette provision (Baseline vs.week 4)
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | NJOY ACE E-cigarette Provision
Number analyzed (Participants) | 15
ppm
  Baseline | 19.4 (11.0)
  Week 4 | 12.3 (8.55)

4. Secondary Outcome: Cigarettes Smoked Per Day After E-cigarette Provision Ends
Description: Self-reported number of cigarettes smoked per day in the past week between end of e-cigarette provision and end of study (week 4 to week 8)
Time Frame: 4 weeks (Weeks 4-8)
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | NJOY ACE E-cigarette Provision
Number analyzed (Participants) | 14
cigarettes/day
  Week 4 | 10.2 (7.0)
  Week 8 | 9.7 (8.0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 8 weeks
Description: Adverse event collection occurred at the end of every study visit using a form where participants were asked about serious adverse events since the previous visit.
Arm/Group | NJOY ACE E-cigarette Provision
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 3/15
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NJOY ACE E-cigarette Provision (N=15)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1
Dizziness or headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT06472869/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT06472869/ICF_001.pdf